CLINICAL TRIAL: NCT00613496
Title: Impact of Irbesartan on Oxidative Stress and C-Reactive Protein Levels in Patients With Persistent Atrial Fibrillation
Brief Title: Irbesartan and Adhesion Molecules in AF
Acronym: CREATIVE-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Magdeburg (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Andreas Goette, MD, University Hospital Magdeburg
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG-1-2007; EUDRACTN: 2007-003262-17
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; irbesartan; AT-II-antagonist; Adhesion Molecules; oxidative stress markers; hsCRP; ICAM; VCAM; MCP-1; vWF; TGFβ1; TNF-α; Interleukin-6; 8isoProstaglandinF2α
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Placebo treatment in each patient during the study (9 weeks) using an intraindividual cross-over design
  Interventions: Drug: placebo
- 1 (Active Comparator): Irbesartan treatment in each patient during the study (9 weeks) using an intraindividual cross-over design
  Interventions: Drug: irbesartan

INTERVENTIONS:
Drug: irbesartan — Irbesartan-tablet (150 mg) 1 in the morning for 7 days, 2 tablets (1 in the morning and 1 in the evening) after day 8 if no contraindication for up titration (investigator will decide on the basis of creatinin, urea and potassium after taking a blood sample) for 9 weeks.
  Other Names: Avapro; Aprovel; Carvea
  Arms: 1
Drug: placebo — Placebo-tablet, 1 in the morning for 7 days, 2 tablets (1 in the morning and 1 in the evening) after day 8.
  Arms: 2

SUMMARY:
Experimental data suggest that angiotensin II-antagonists reduce the atrial expression of prothrombotic adhesion molecules and oxidative stress parameters. The present study is designed to investigate the effects on angiotensin II-antagonist irbesartan to reduce the amounts of circulating oxidative stress markers and adhesion molecules in patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
Primary Objective:

The aim of the study is to assess that blocking the angiotensin II type 1 receptor reduces systemic levels of oxidative stress markers and adhesion molecules by more than 25% compared to placebo in patients with persistent/permanent atrial fibrillation.

Primary Target Parameter:

The primary target parameter is defined as reduction of systemic levels of oxidative stress markers and adhesion molecules (hsCRP, ICAM, VCAM, MCP-1, vWF, TGFβ1, TNF-α, Interleukin-6, 8isoProstaglandinF2α)

Secondary Target Parameter:

The secondary Target Parameters are defined as number of cerebrovascular events, number of intermediate medical visits for cardiovascular reasons without hospitalisation, number of hospitalisations for cardiovascular reasons and GFR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent/permanent AF (>2 months)
* CHADS2 Score ≥2
* Age ≥18
* Patient informed orally and in writing
* Written informed consent of the patient
* Patients who are anticipated to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 148 days clinical follow-up
* Patients who are mentally and linguistically able to understand the aim of the study and the associated risks and benefits of the treatment. The patients, by providing informed consent, agree to this treatment as stated in the patient informed consent document.

Exclusion Criteria:

* Strong clinical evidence that prevents the temporary pause of therapy with AT II antagonists
* Symptomatic bradycardia
* Implanted pacemaker or implanted cardioverter/defibrillator with any antitachycardia algorithm in use
* Cardiac surgery or cardiac catheter ablation within the last 3 months prior to randomisation
* Typical angina pectoris symptoms at rest or during exercise
* Known coronary artery disease with indication for intervention
* Symptomatic peripheral vascular disease
* Left ventricular ejection fraction <35%
* Myocardial infarction within 6 months prior to randomisation
* Diastolic blood pressure >110mmHg at rest
* Symptomatic arterial hypotension
* Known renal artery stenosis
* Serum creatinin >1.8mval/l
* Chronic inflammatory disease
* Acute inflammatory disease (CRP >20mg/L)
* Relevant hepatic or pulmonary disorders
* Hyperthyreosis manifested clinically and in laboratory
* Known drug intolerance for AT II inhibitors
* Females who are pregnant or breast feeding
* Females of childbearing potential who are not using a scientifically accepted method of contraception
* Participation in a clinical trial within the last 30 days prior to randomisation
* Drug addiction or chronic alcohol abuse
* Cancer or other disease, which inevitably leads to death
* Legal incapacity, or other circumstances which would prevent the patient from understanding the aim, nature or extent of the clinical study, evidence of an uncooperative attitude

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The primary target parameter is defined as reduction of systemic levels of oxidative stress markers and adhesion molecules (hsCRP, ICAM, VCAM, MCP-1, vWF, TGFβ1, TNF-α, Interleukin-6, 8isoProstaglandinF2α) | 22 weeks

SECONDARY OUTCOMES:
Number of cerebrovascular events | 22 weeks
Number of intermediate medical visits for cardiovascular reasons without hospitalization | 22 weeks
Number of hospitalization for cardiovascular reasons and GFR | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Goette, MD, Principal Investigator — University Hospital Magdeburg; Div of Cardiology
Locations (1):
- University Hospital Magdeburg; Div. of Cardiology, Magdeburg, Germany